CLINICAL TRIAL: NCT02137486
Title: Outcome of Coronary High Angulated Bifurcation Lesions Treated With Kissing Ballooning or Sequential Ballooning Techniques
Acronym: MV:main branch
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Yueh-Chung, Chen, chief of ICU, Taipei City Hospital
Other Study IDs: TCHIRB-1030209-E
Record Dates: First submitted 2014-04-19; First posted 2014-05-13 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2017-04

CONDITIONS: Stable Angina
Keywords: stable angina; high angulated bifurcation; SYNTAX; DES; BMS
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sequential ballooning: include BMS or DES
- final kissing ballooning: include BMS or DES

SUMMARY:
Coronary artery bifurcation lesions prone to occur with the worsening of atherosclerosis. Their structural properties make angioplasty technique to increase the difficulty of implementation, but also increased the risks of the in-stent thrombosis and restenosis. Standard treatment of coronary bifurcation lesions remains controversial manner, especially when the side branch (SB) was large combined with high angulated bifurcation lesions. Complex procedures and certain types of lesions are associated with poor prognosis. There is no standard treatment for such lesions even with the development of drug-eluting stents solve partial problems. The investigators reviewed patients who received coronary intervention between 2009-2012 years and met the inclusion criteria, and then analyzed the prognostic relevance of these cases the use of different treatment modalities.

We introduced a retrospective analysis for high angulated bifurcation lesions treated with either DES or BMS.

Primary endpoint: cardiovascular mortality, TLR, MACE. secondary endpoint: procedure time, fluoroscopy time, procedure success, angiographic success.

ELIGIBILITY:
Inclusion Criteria:

* Angulated bifurcation:MV(main branch) and SB(side branch) angle>70 degree. MV diameter≥2.5mm and eligible for stenting. lesion stenotic severity>70% by QCA(Quantitative coronary analysis). 1 stent strategy. SYNTAX>22 Procedure success. de novo lesion

Exclusion Criteria:

* Bifurcation lesions intervention without side br. ballooning after stents deployment or procedure incomplete. Left main coronary artery bifurcational lesions. Elective,provisional or bail-out stenting for side br.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients revceived coronary intervention between 2009-2014/3.
Sampling Method: Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei city hospital, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequential Ballooning: the stent is placed in the MV and dilated, and then a second balloon just proximal to the opening of the SB is dilated in order to widen the diameter of the MV at the SV opening to allow more blood to be diverted into the SB; then treated with drug eluting stent or bare metal stent.
- Final Kissing Ballooning: a balloon that extends from a position in the MV just proximal to the SB into a portion of the SB is inflated at the same time as the MV balloon; then treated with drug eluting stent or bare metal stent.
Period: Overall Study
Arm/Group | Sequential Ballooning | Final Kissing Ballooning
Started | 112 | 102
Completed | 112 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: high angle bifurcation lesion
Groups:
- Sequential Ballooning; Final Kissing Ballooning: treated with drug eluting stent or bare metal stent.
- Total: Total of all reporting groups
Arm/Group | Sequential Ballooning | Final Kissing Ballooning | Total
Number analyzed (Participants) | 112 | 102 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 78 | 160
  >=65 years | 30 | 24 | 54
Age, Continuous [Median (Standard Deviation); unit: years] | 68.69 (11.43) | 67.67 (11.49) | 67.98 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 87 | 81 | 168
Region of Enrollment [Number; unit: participants]
  Taiwan | 112 | 102 | 214

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Adverse Cardiac Events(MACE)
Description: Percentage of Participants with major adverse cardiac events(MACE) was defined as rates of target lesion revascularization (TLR) and restenosis during first post-treatment year, and rates of acute, subacute, and late in-stent thrombosis, periprocedure MI(myocardial infarction).
Time Frame: periprocedure up to 12 months
Population: 100%x2/112; 100%x7/102
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sequential Ballooning | Final Kissing Ballooning
Number analyzed (Participants) | 112 | 102
percentage of participants | 1.72 [1.24 to 1.98] | 6.86 [6.01 to 7.14]

2. Primary Outcome: Percentage of Participants With Cardiovascular Mortality(%)
Description: Percentage of Participants with cardiovascular mortality was defined as death related to cardiovascular causes within 2 years.
Time Frame: periprocedure up to 12 months
Population: 100%x0/112; 100%x1/102
Measure: Count of Participants; unit: Participants
Arm/Group | Sequential Ballooning | Final Kissing Ballooning
Number analyzed (Participants) | 112 | 102
Participants | 0 | 1

3. Secondary Outcome: Percentage of Participants With Angiographic Success(%)
Description: Percentage of Participants with angiographic success was defined as residual stenosis<50% under fluoroscopy at the end of procedure.
Time Frame: periprocedure up to 12 months.
Population: lesions of participants; 100%x90/112; 100%x84/102.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequential Ballooning | Final Kissing Ballooning
Number analyzed (Participants) | 112 | 102
Participants | 90 | 84

4. Secondary Outcome: Percentage of Participants With Target Vessel Revascularization Rate
Description: Percentage of Participants with target vessel revascularization rate, both arms
Time Frame: periprocedure up to 12 months.
Population: Percentage of Participants with target vessel revascularization rate, both arms
Measure: Count of Participants; unit: Participants
Arm/Group | Sequential Ballooning | Final Kissing Ballooning
Number analyzed (Participants) | 112 | 102
Participants | 24 | 19

5. Secondary Outcome: Fluoroscopy Time(Minutes) of Each Participants
Description: as medical chart record.
Time Frame: periprocedure up to 12 months.
Population: fluoroscopy time(minutes) of each participants
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sequential Ballooning | Final Kissing Ballooning
Number analyzed (Participants) | 112 | 102
minutes | 24 (6) | 36 (4)

6. Secondary Outcome: Procedure Time(Minutes) of Each Participants
Description: as medical chart record.
Time Frame: periprocedure up to 12 months.
Population: procedure time(minutes) of each participants
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sequential Ballooning | Final Kissing Ballooning
Number analyzed (Participants) | 112 | 102
minutes | 84 (8) | 92 (4)

ADVERSE EVENTS:
Arm/Group | Sequential Ballooning | Final Kissing Ballooning
All-Cause Mortality (participants affected / at risk) | 0/112 | 1/102
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/102
Other Adverse Events (participants affected / at risk) | 0/112 | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes